CLINICAL TRIAL: NCT01426451
Title: Assessment of a Drama Workshop Program for Immigrant and Refugee Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Cécile Rousseau, Associate Professor, Division of Social and Cultural Psychiatry, McGill University, Transcultural Research and Intervention Team (TRIT), Youth Mental Health, CSSS de la Montagne (Park Extension), McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIHR/IRSC-229984
Record Dates: First submitted 2011-08-25; First posted 2011-08-31 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Learning Disabilities
Keywords: Dramatherapy; Group tutoring activities; Impairment; Emotional and behavioural problems; Learning difficulties
MeSH Terms: conditions — Learning Disabilities; Mental Disorders

ARMS (3):
- Theatre intervention (Experimental): The theatre expression workshops will run for 12 weeks, with one 75-minute workshop per week. They will be incorporated into the regular class timetable and will be run by the two members of the intervention team who have training in theatre and psychology, and the homeroom teacher, whose level of direct involvement will increase gradually as he or she becomes familiar with the workshops.
  Interventions: Other: Theatre workshops
- Group tutoring intervention (Experimental): In each classroom assigned to the tutorship intervention, two academic resource assistants will provide weekly in-class support to students for the same length of time than the drama workshop (75 minutes weekly). Individualized student objectives on reading fluency and math will be implemented (one in math and one in reading per student).
  Interventions: Other: Group tutoring program
- No intervention (No Intervention): Classes not participating neither in drama workshops nor in group tutoring activities will fill out a questionnaire as a basis for comparison.

INTERVENTIONS:
Other: Group tutoring program — Academic in-class intervention that focuses on differentiated academic instruction and improved overall academic adjustment. In each classroom assigned to the tutorship intervention, two academic resource assistants will provide weekly in-class support to students for the same length of time than the drama workshop (75 minutes, once a week), with the teacher present in the classroom.
  Arms: Group tutoring intervention
Other: Theatre workshops — The theatre expression workshops will run for 12 weeks, with one 75-minute workshop per week. They will be incorporated into the regular class timetable and will be run by the two members of the intervention team who have training in theatre and psychology, and the homeroom teacher, whose level of direct involvement will increase gradually as he or she becomes familiar with the workshops.
  Arms: Theatre intervention

SUMMARY:
The purpose of this study is to determine whether a drama workshop program for immigrant and refugee youth is effective in reducing impairment in high school students presenting learning difficulties.

ELIGIBILITY:
Inclusion Criteria:

* All students who are assigned to special classes based on behavioural or learning problems in grades 7-10 in the participating schools will participate in the program and be included in the study if they and their parents consent to in the research.

Exclusion Criteria:

* More severe cases

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 464 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in impairment of emotional and behavioural symptoms reported by youth | T0: up to 6 weeks before the intervention, T1: up to 2 weeks after the intervention, T2: between 7 and 8 months after the intervention
  Impairment of emotional and behavioural symptoms will be assessed by the Impact Supplement of the SDQ completed by the adolescents. The SDQ is a 25-item Likert scale assessing emotional and behavioural symptoms. This questionnaire includes an impairment measure that enquires about symptoms in terms of chronicity, distress, social impairment, and burden for others.

SECONDARY OUTCOMES:
Change in emotional and behavioural symptoms | T0: up to 6 weeks before the intervention, T1: up to 2 weeks after the intervention, T2: between 7 and 8 months after the intervention
  Will be assessed by the SDQ global scores (teachers and youths reports).
Change in impairment | T0: up to 6 weeks before the intervention, T1: up to 2 weeks after the intervention, T2: between 7 and 8 months after the intervention
  Measured by the SDQ (teacher report).
Change in relations with peers | T0: up to 6 weeks before the intervention, T1: up to 2 weeks after the intervention, T2: between 7 and 8 months after the intervention
  Will be assessed using the Adolescent Friendship Inventory (AFI) designed by Rubenstein et al. (1989). This 30-item instrument requires the adolescent to indicate to what degree, on a scale of 1 to 5, the feeling expressed by the statement corresponds to his or her personal feelings in relation to his or her network of peers.
Change in school performance | T0: up to 6 weeks before the intervention, T1: up to 2 weeks after the intervention, T2: between 7 and 8 months after the intervention
  Will be assessed on the basis of the first and the last report cards of the school year (T0 and T1) and with the first report card of the subsequent year (T2). We will consider students' grades in mathematics and French.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Rousseau, MD, Principal Investigator — McGill University Health Center, CSSS de la Montagne
Locations (5):
- Canada (5):
  - École Antoine-de-St-Exupéry, Montreal, Quebec
  - École La Dauversière, Montreal, Quebec
  - École La Voie, Montreal, Quebec
  - École Lucien-Pagé, Montreal, Quebec
  - École Saint-Luc, Montreal, Quebec

REFERENCES:
- [Derived] Rousseau C, Beauregard C, Daignault K, Petrakos H, Thombs BD, Steele R, Vasiliadis HM, Hechtman L. A cluster randomized-controlled trial of a classroom-based drama workshop program to improve mental health outcomes among immigrant and refugee youth in special classes. PLoS One. 2014 Aug 15;9(8):e104704. doi: 10.1371/journal.pone.0104704. eCollection 2014. PMID 25127251